CLINICAL TRIAL: NCT07333417
Title: The Effect of Rigid Taping on Pain and Function in Individuals With Acromioclavicular Joint
Brief Title: Effects of Rigid Taping in Acromioclavicular Joint Degeneration
Acronym: ACJTaping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, Professor, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACJTaping
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain; Acromioclavicular Joint
Keywords: Shoulder pain; Acromioclavicular joint degeneration; Rigid taping
MeSH Terms: conditions — Shoulder Pain | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Outcome assessments are planned to be conducted by an assessor blinded to group allocation whenever possible.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rigid Taping + Exercise (Active Comparator): Participants will receive rigid acromioclavicular joint taping once weekly for 4 weeks in addition to a standardized shoulder exercise program supervised by a physiotherapist.
  Interventions: Other: Rigid Taping; Other: Exercise Program
- Exercise Only (Active Comparator): Participants will receive a standardized shoulder exercise program supervised by a physiotherapist without any taping application.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Rigid Taping — Rigid taping will be applied to the acromioclavicular joint using a standardized technique aiming to posteriorize the acromion and inferiorize the clavicle. Taping will be performed once weekly for 4
  Arms: Rigid Taping + Exercise
Other: Exercise Program — A standardized shoulder exercise program focusing on soft tissue flexibility, scapular stabilization, and rotator cuff activation will be applied once weekly for 4 weeks.

SUMMARY:
This study will examine whether rigid taping applied to the acromioclavicular (AC) joint can reduce shoulder pain and improve shoulder function in people with AC joint degeneration. Participants with shoulder pain and a confirmed diagnosis of AC joint degeneration will be randomly assigned to one of two groups: (1) rigid taping plus a standardized exercise program or (2) the same exercise program without taping. The program will last 4 weeks, with weekly supervised visits. Pain, shoulder motion, and shoulder function will be assessed at baseline, after the first session (acute effect), at the end of treatment (Week 4), and at a 3-month follow-up.

DETAILED DESCRIPTION:
Shoulder pain is one of the most common musculoskeletal complaints and can affect daily activities, work, and sports participation. Among the potential sources of shoulder pain, the acromioclavicular (AC) joint is a distinct pain generator that can often be identified through a targeted clinical examination. Diagnosis is typically based on a detailed history combined with physical tests designed to provoke AC joint symptoms, such as scarf maneuvers and localized palpation.

The AC joint is a synovial articulation between the distal clavicle and the acromion of the scapula. Although its motion is relatively limited, it plays an important role in load transfer across the shoulder girdle, particularly during arm elevation and overhead activities. AC joint symptoms may arise through different mechanisms, including degenerative changes over time, traumatic events, or inflammatory processes. Degenerative AC joint disease may coexist with other shoulder conditions, and structural changes around the joint can contribute to pain by increasing mechanical stress and altering the subacromial environment. As a result, individuals may experience pain with overhead movements, cross-body motions, lifting, pushing, or during sport-specific tasks.

Management of AC joint degeneration typically begins with conservative care. Common non-surgical strategies include physiotherapy, activity modification, temporary unloading or immobilization when needed, and symptom-directed medical management. Rehabilitation approaches generally focus on optimizing posture, improving scapular control, enhancing periscapular strength and endurance, restoring flexibility of the posterior shoulder structures, and progressively reintroducing functional loading while minimizing symptom provocation.

Taping techniques are frequently used in shoulder rehabilitation as an adjunct to exercise-based care. In clinical practice, rigid and elastic taping methods are applied with the intention of modifying joint alignment and mechanical loading, limiting painful movement patterns, and supporting more efficient scapulothoracic and glenohumeral mechanics during activity. Rigid taping, in particular, is often considered when a more structured mechanical effect is desired. While taping has been investigated in various shoulder pain presentations, existing evidence has largely focused on subacromial pain conditions and scapular kinematics rather than AC joint degeneration specifically. Consequently, there remains uncertainty about whether rigid taping provides additional clinical benefit for individuals whose primary pain source is degenerative change at the AC joint.

Therefore, the purpose of this study is to evaluate the effects of rigid AC joint taping on shoulder pain, pain-free shoulder range of motion, and shoulder function in individuals with shoulder pain associated with AC joint degeneration.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of acromioclavicular (AC) joint degeneration confirmed by clinical examination and imaging (X-ray, ultrasound, or MRI).
* Shoulder pain duration of at least 4 weeks.
* Age between 18 and 65 years
* Willingness to refrain from any additional treatments outside the study protocol during the study period (e.g., medication changes, injections, or physiotherapy elsewhere) and to provide written informed consent

Exclusion Criteria:

* Current or previous diagnosis/history of acromioclavicular (AC) joint separation.
* Diagnosis of frozen shoulder (adhesive capsulitis).
* History of acute trauma or fracture involving the shoulder girdle (e.g., clavicle fracture, shoulder dislocation).
* History of shoulder surgery.
* Systemic inflammatory joint disease (e.g., rheumatoid arthritis) or other systemic arthropathies.
* Skin conditions preventing taping (e.g., rash, open wound, or known tape allergy).
* Neuromuscular disease or neurological disorders affecting shoulder function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (Week 0), immediately after the first session (acute effect), Week 4 (end of intervention), and Month 3 follow-up
  Pain intensity will be assessed at rest and during activity using the Visual Analog Scale (VAS).
Shoulder Range of Motion | Baseline (Week 0), immediately after the first session (acute effect), Week 2, Week 4 (end of intervention), and Month 3 follow-up
  Shoulder range of motion (flexion, abduction, internal rotation, and external rotation) will be assessed using a goniometer by recording active range of motion until pain onset, active range of motion despite pain, and passive end-range of motion.

SECONDARY OUTCOMES:
Shoulder Function | Baseline (Week 0), Week 4 (end of intervention), and Month 3 follow-up
  Shoulder function will be evaluated using the American Shoulder and Elbow Surgeons Shoulder Score (ASES), which assesses pain and functional activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Sports Physiotherapy and Rehabilitation Department, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because specific data-sharing agreements and governance procedures have not been established.